CLINICAL TRIAL: NCT06353230
Title: Comparison of Sclerotherapy Agents Used for Rectal Prolapse Treatment in Children
Acronym: Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Muhammad Sharif, PROFESSOR, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2024-03-31; First posted 2024-04-09 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Rectal Prolapse
Keywords: Injection Sclerotherapy; 5% Phenol in Almond oil; 15%Hypertonic saline; 50% dextrose water; Rectal prolapse
MeSH Terms: conditions — Rectal Prolapse | interventions — Injections; Phenol; almond oil; Saline Solution, Hypertonic; Sclerotherapy

STUDY DESIGN:
Intervention Model Description: Comparison of 5% phenol in almond oil, 15% hypertonic saline and 50% dextrose water for sclerotherapy treatment of rectal prolapse in children.
Masking Description: Randomly allocated groupA,B or C by computer generated lottery method.and participants ,care provider and outcome assessor were kept blind by removing the drug name from injection vial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A with 5% phenol in almond oil (Experimental): Group A patients with rectal prolapse were given injection sclerotherapy with 5% phenol in almond oil,
  Interventions: Procedure: injection 5% phenol in almond oil; Procedure: injection 15% hypertonic saline; Procedure: injection 50% dextrose water
- Group B with hypertonic saline (Active Comparator): Group B with rectal prolapse were given injection sclerotherapy with 15% hypertonic saline
  Interventions: Procedure: injection 5% phenol in almond oil; Procedure: injection 15% hypertonic saline; Procedure: injection 50% dextrose water
- Group C with 50% Dextrose water (Active Comparator): Group C with rectal prolapse were given injection sclerotherapy with 50% Dextrose water
  Interventions: Procedure: injection 5% phenol in almond oil; Procedure: injection 15% hypertonic saline; Procedure: injection 50% dextrose water

INTERVENTIONS:
Procedure: injection 5% phenol in almond oil — Group A were given 5% phenol in almond oil
  Other Names: sclerotherapy wiyh 5% phenol in almond oil
Procedure: injection 15% hypertonic saline — Group B were given hypertonic saline
  Other Names: sclerotherapy with hypertonic saline
Procedure: injection 50% dextrose water — group C were given 50% dextrose water
  Other Names: sclerotherapy with 50% dexrose water

SUMMARY:
Introduction Patients with rectal prolapse are treated with injection sclerotherapy, which is the most often used first-line surgical technique. Injection sclerotherapy has a success rate of 90-100% in youngsters, according to certain studies. Objective To compare the outcome of injection sclerotherapy using 5% Phenol in almond oil, 15% hypertonic saline and 50% dextrose water in the treatment of rectal prolapse in children.

DETAILED DESCRIPTION:
Materials and Methods Study design: Randomized control trial. Setting: Paediatric surgery department, King Edward medical university, Mayo Hospital Lahore. Duration: Twelve months after approval of synopsis. Data collection procedure: After ethical approval, all the patients with rectal prolapse fulfilling inclusion criteria admitted. Routine history, thorough clinical examination and routine preoperative investigations was done. Patients were randomly allocated to group A, B or C using the lottery method. Group A patients were given injection sclerotherapy with 5% phenol in almond oil; Group B patients were given injection sclerotherapy with 15% hypertonic saline and group C patients were given injection sclerotherapy with 50% dextrose water solution. Under general anesthesia and patient in lithotomy position, 2-3 ml of sclerosing agent was injected into the submucosa at 3 sites around the circumference preferably at 3,6 and 9'o' clock positions about 2-3 cm above dentate line. The injection was performed under vision, using a speculum while LP needle was passed through the perianal skin. All patients were kept under observation during the hospital stay and discharged on same day and followed on week 1 and after 3 months for recurrence of rectal prolapse, fecal incontinence, perianal abscess and anal stenosis according to the operational definition.

ELIGIBILITY:
Inclusion Criteria:

• Patients with partial or complete rectal prolapse of either gender presenting to paediatric surgery department, Mayo Hospital Lahore, under 13 years of age.

Exclusion Criteria:

* Patients of rectal prolapse due to ulcerative colitis and crohn's disease documented in medical record.
* Patients with previous history of surgery on pelvic floor documented in medical record.
* Caudaequina syndrome, neural tube defects, Sacrococcygeal teratoma, Hirschsprung,s disease, congenitalmega colon and rectal polyps documented in medical record. -

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
Recurrence | 3 months
  Re-appearance of signs and symptoms of rectal prolapse after remission will be labelled as

SECONDARY OUTCOMES:
fecal incontinence | 3 months
  Kelly Score will be used to assess fecal incontinence. Kelly score includes 3 parameters; occurrence of accidents, soiling and anal sphincter action. Each parameter will be scored between 0-2 with total score of 6. Total score 5 or 6 will be labelled as good fecal continence, 3 or 4 score is fair and 0 to 2 score will be labelled as poor fecal continence

CONTACTS AND LOCATIONS:
Locations (1):
- department of pediatric surgery King Edward Medical University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Will be shared through personal request